CLINICAL TRIAL: NCT02710240
Title: A Pilot/Feasibility Study of Intraoperative Image-Guided Surgery of CNS Tumors With Indocyanine Green and MR Spectroscopic Imaging
Brief Title: Indocyanine Green for Central Nervous System Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPCC 09315
Record Dates: First submitted 2016-03-14; First posted 2016-03-16 (Estimated); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Suspected Central Nervous System Tumors
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICG Arm (Experimental): Subjects undergo indocyanine green injection within 72 hours prior to surgery. Permitting infusion time within 72 hours of operation is believed to be adequate for tissue glow/surgical visualization. Alternately, patients may receive 25 mg of indocyanine green during induction. Dose and time of administration will be determined by the neurosurgeon during surgical planning. This 25 mg dose of indocyanine green is similar to dosing for other intraoperative vascular visualization.
  Interventions: Drug: Indocyanine Green (ICG); Radiation: Intraoperative near-infrared (NIR)

INTERVENTIONS:
Drug: Indocyanine Green (ICG)
Radiation: Intraoperative near-infrared (NIR)

SUMMARY:
This study is a single center, open-label, two-part study to assess image guided surgery of intramolecular imaging in nervous system tumors. Subjects with a diagnosis of a resectable nervous system tumor who are at risk of recurrence are included. The primary goal is to observe what tissues fluoresce in the OR, and then to identify if that tissue is cancerous/tumor or normal when the histopathology is performed.

ELIGIBILITY:
Inclusion Criteria:

Adult patients 18 years of age and older Patients presenting with a CNS tumor presumed to be resectable and are at risk for local recurrence on pre-operative assessment Good operative candidate as determined by the treating physician and multidisciplinary team Subject capable of giving informed consent and participating in the process of consent

Exclusion Criteria:

Pregnant women as determined by urinary or serum beta hCG within 72 hours of surgery Subjects with a history of iodide allergies Vulnerable patient populations Patients unable to participate in the consent process (children and neonates) Patients with non-MRI compatible implanted metallic foreign bodies Patients who due to severe claustrophobia cannot tolerate MRI scanning Patients with a known allergy or hypersensitivity to MRI contrast agents including gadolinium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lee, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Cho SS, Sheikh S, Teng CW, Georges J, Yang AI, De Ravin E, Buch L, Li C, Singh Y, Appelt D, Delikatny EJ, Petersson EJ, Tsourkas A, Dorsey J, Singhal S, Lee JYK. Evaluation of Diagnostic Accuracy Following the Coadministration of Delta-Aminolevulinic Acid and Second Window Indocyanine Green in Rodent and Human Glioblastomas. Mol Imaging Biol. 2020 Oct;22(5):1266-1279. doi: 10.1007/s11307-020-01504-w. PMID 32514886

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ICG Arm
Started | 336
Completed | 336
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ICG Arm
Number analyzed (Participants) | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191
  Male | 145
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 336

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity (SBR)
Description: sensitivity of delayed, high dose indocyanine green (second window ICG), as measured by the signal-to-background ratio (SBR)
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ICG Arm
Number analyzed (Participants) | 336
ratio | 5.49 (3.20)

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | ICG Arm
All-Cause Mortality (participants affected / at risk) | 118/336
Serious Adverse Events (participants affected / at risk) | 3/336
Other Adverse Events (participants affected / at risk) | 13/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICG Arm (N=336)
Hypertension (Cardiac disorders) | 3 (3) — 1. patient experienced hypertension pre-infusion. 2. patients experienced from hypertension during infusion and infusion was discontinued. These events were classified as SAEs as the patients were taken to the ED for treatment.
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 patient experienced respiratory distress during infusion and infusion was discontinued.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ICG Arm (N=336)
IV Site Reactions (Skin and subcutaneous tissue disorders) | 4 (4) — 4 patients experienced IV site reactions during infusion. No treatment was deemed necessary and patients recovered upon observation.
Hypertension (Cardiac disorders) | 3 (3) — 3 patients experienced hypertension during infusion. Infusion was stopped for 1 patient. Infusion was slowed and completed for 1 patient. No action was taken for 1 patient. Hypertension resolved for all 3 patients upon observation.
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 patient experienced hypoxia post-infusion. No treatment was deemed necessary. O2 levels recovered in time upon observation.
Itching (Skin and subcutaneous tissue disorders) | 2 (2) — 2 patients experienced itching during infusion. Both patients received Benadryl, after which the itching resolved.
Hives (Skin and subcutaneous tissue disorders) | 1 (1) — 1 patient experienced hives during infusion. The patient received Benadryl, after which the hives resolved.
Foot Drop (Musculoskeletal and connective tissue disorders) | 1 (1) — 1 patient experienced foot drop, presumed secondary to brain tumor. AE was determined to be unrelated and unexpected by the study investigator.
Nausea (Gastrointestinal disorders) | 1 (1) — 1 patient reported nausea during infusion. Infusion was discontinued and the symptoms resolved.
Vomiting (Gastrointestinal disorders) | 1 (1) — 1 patient began to vomit during infusion. Infusion was discontinued and the symptoms resolved.
Unilateral Upper Extremity Pain (Musculoskeletal and connective tissue disorders) | 2 (2) — 2 patients reported upper extremity pain on the side of the IV placement and infusion. Infusion was discontinued for 1 patient and symptoms resolved. No action was taken for 1 patient and symptoms resolved upon observation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT02710240/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT02710240/ICF_001.pdf